CLINICAL TRIAL: NCT06945731
Title: The Effectiveness of Repetitive Transcranial Magnetic Stimulation for Weight Loss in Overweight and Obese Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Nikolaos Liaskopoulos, MD, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28/01/2022/3672
Record Dates: First submitted 2025-04-01; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Obesity and Overweight; Food Cravings
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator)
  Interventions: Device: TMS
- Sham (Sham Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: TMS — 20 sessions 10 Hz rTMS
  Arms: Active
Device: Transcranial Magnetic Stimulation Sham — Sham TMS
  Arms: Sham

SUMMARY:
This doctoral dissertation takes into account epidemiological and clinical data of the international literature about obesity and, generally, increased body weight (BMI≥ 25kg/m2) and their consequences on health. Obesity management challenges many specialties, while, currently, the approved therapeutic methods are dietary intervention, various drugs and, in severe cases, bariatric surgery. All of the above methods show some degree of recurrence, while surgery carries the risk of serious complications.

Repetitive transcranial magnetic stimulation (rTMS) is classified into non-invasive brain stimulation methods and utilizes magnetic pulses generated by a coil to bring about changes in the brain. The method has already been approved for the treatment of some disorders, while it seems to help in the fight against many more psychiatric and neurological, mainly, diseases. The aim of the research will be to investigate the effectiveness of TMS in reducing body weight in participants with BMI≥ 25kg/m2.

The doctoral dissertation will study the reduction of BMI in obese and overweight patients and the variation of this reduction depending on the severity of obesity and age. In addition, it will investigate the effectiveness by setting as a parameter the observance of a diet. It will also record and statistically process the improvement of symptoms in the spectrum of some psychiatric disorders (eg depressive and psychotic symptoms, psychosomatic disorders).

The participants in the research will be hospitalized patients of the Psychiatric Clinic of the University General Hospital of Larissa (PGNL) and citizens. Clearly, patients from other clinics or other citizens can also participate in the research, provided they have a BMI≥ 25kg/m2. They will undergo 20 rTMS sessions (4 per week, for 5 weeks) and an assessment of BMI and some psychiatric symptoms before the start, at the end, 4 weeks after and 6 months after the end of the sessions. The rTMS will be applied to the left dorsal prefrontal cortex (left DLPFC), with an 8-coil in the following conditions: frequency 10 Hz, 75 4-second trains with 26-second intertrain interval, at 120% of the threshold for motor cortex activation. Participants will be divided into three groups: those who will not receive TMS, those who will receive sham TMS and those who will receive active TMS. These patients will then be compared with each other to answer the research questions. The therapeutic protocol presented is based on the international literature, while it presents positive results in the studies in which it has been applied.

Prerequisites for participation in the study are patient consent and BMI≥ 25kg/m2. In order to receive TMS, the patient first needs to agree and clarify that he / she does not have an individual or family history of seizures and that he / she does not have a cochlear implant. If the patient wishes, he can withdraw from the study at any stage. In addition to seizures, other side effects of treatment include headache and hearing loss (for which the patient will use earplugs).

The present dissertation will contribute to the further understanding of the mechanisms of obesity as well as the development of new therapies for the treatment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* BMI > 25 kg/m²
* Ability to provide written consent

Exclusion Criteria:

* History of epilepsy
* Active alcohol or substance abuse
* Severe active health condition
* Cochlear implants
* Inability to provide written consent
* BMI < 25 kg/m²
* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-28 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
BMI | From enrollment to the end of the treatment at 5 weeks, follow up of 1 month and 6 months
Food Craving | From enrollment to the end of the treatment at 5 weeks, follow up of 1 month and 6 months
  Scale: Food Cravings Questionnaire-Trait Scores: 15-90 Higher score means worsening of symptoms

SECONDARY OUTCOMES:
Depressive Symptoms | From enrollment to the end of the treatment at 5 weeks, follow up of 1 month and 6 months
  Scale Patient Health Questionnaire 9 Scores 0-27 Higher Score means worsening of symptoms
Anxiety symptoms | From enrollment to the end of the treatment at 5 weeks, follow up of 1 month and 6 months
  Generalised Anxiety Disorder Questionnaire 7 Scores 0-21 Higher Score means worsening of symptoms
Psychosomatic symptoms | From enrollment to the end of the treatment at 5 weeks, follow up of 1 month and 6 months
  Scale Patient Health Questionnaire 15 Scores 0-30 Higher Score means worsening of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Universital General Hospital of Larissa, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No